CLINICAL TRIAL: NCT03276520
Title: Filling the Gap Between Lab and Clinical Impact: an Open Randomized Diagnostic Trial Comparing Urinary Ethylglucuronide and Ethanol in Alcohol Dependent Outpatients.
Brief Title: Randomized Diagnostic Trial Comparing Ethylglucuronide and Ethanol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Antoni Gual, Head of Addictive Behaviors Unit, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HCB/2015/0984
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Alcohol Use Disorder
Keywords: ethyl glucuronide, biomarker, diagnostic randomized trial
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ethyl glucuronide (Experimental): subjects being screened with ethyl glucuronide
  Interventions: Diagnostic Test: ethyl glucuronide
- ethanol (Active Comparator): subjects being screened with ethanol
  Interventions: Diagnostic Test: ethanol

INTERVENTIONS:
Diagnostic Test: ethyl glucuronide — alcohol urine screening with ethyl glucuronide
  Arms: ethyl glucuronide
Diagnostic Test: ethanol — alcohol urine screening with ethanol
  Arms: ethanol

SUMMARY:
Background: Alcohol use disorders represent a major health burden. Efforts aiming at reducing alcohol-related harm include early detection of those with risky drinking habits as well detection of early relapse in patients with alcohol dependence who are detoxified and committed to abstinence. Recently, ethyl glucuronide has been proved to be a good biomarker for the detection of recent drinking. However, to date, no randomized diagnostic trial has tested its impact on drinking outcomes. The aim of this study was to assess, with a randomized design, the implications of ethyl glucuronide screening on alcohol outcomes, compared to screening with a low-sensitivity biomarker such as ethanol.

Methods: alcohol dependent outpatients were randomized to either 24 weeks of continuous screening with ethyl glucuronide or ethanol. Patients were aware of screening methods and results. After 24 weeks, all participants were screened with ethyl glucuronide. Self-reports were also gathered. A logistic regression model was performed comparing the rate of ethyl glucuronide positive results at study end between groups. Generalized estimating equations were performed to evaluate the descending rate of EtG positive patients in the EtG group, measured month to month.

ELIGIBILITY:
Inclusion Criteria:

* subjects had to be diagnosed of alcohol dependence according to DSM-IV, they had to undergo regular urine screening as part of their treatment and be willing to give informed written consent.

Exclusion Criteria:

* conditions rendering patients unable to complete study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
ethyl glucuronide positive rate | after six months of ongoing urine screening
  Percentage of patients screening positive to EtG at study end in each group
descending of Etg positive rates in the Etg group | six months of ongoing urine screening
  varying rate of EtG positive patinets in the intervention group during the study period